CLINICAL TRIAL: NCT03050281
Title: Utility, Feasibility, and Cost-effectiveness of Using a Combined Cadaver and Simulation Laboratory Experience During the OB-GYN and Surgical Medical School Clerkships
Brief Title: Simulation and Cadaver Workshop for Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brian Shapiro, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-003385
Record Dates: First submitted 2016-11-04; First posted 2017-02-10 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Educational Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simulation/Cadaver Workshop (Experimental): 2-day workshop using the Simulation/Cadaver Lab
  Interventions: Other: Simulation/Cadaver lab
- Didactic Workshop (Placebo Comparator): Lectures
  Interventions: Other: Lectures

INTERVENTIONS:
Other: Simulation/Cadaver lab — The primary focus of this study is to determine whether the use of a comprehensive, combined, and simplified approach of using cadavers and simulation laboratories to train third-year medical students will have a beneficial effect on student performance in the OB-GYN and surgical clerkships.
  Arms: Simulation/Cadaver Workshop
Other: Lectures — Standard Anatomy lectures were offered.
  Arms: Didactic Workshop

SUMMARY:
Background: The use of simulation and cadaveric laboratory training are highly beneficial for faculty and advanced trainees, but its usefulness for third-year medical students rotating through OB-GYN or general surgery is unknown.

Objective: To determine if a two-day intensive, cost-effective review of procedural skills and anatomy using the simulation laboratory and cadaver-based dissection improves performance of third-year medical students on the National Board of Medical Examiners (NBME) Shelf and USMLE Step 2 board examination and during pre- and post-test demonstrations.

Significance: If proven effective, implementation of a short, inexpensive, and comprehensive course highlighting anatomical and procedural skills during the third year of medical school could be implemented.

Design Methods: The investigators will conduct a 1:1 randomization of third-year medical students rotating at all Mayo sites (Jacksonville, Rochester, and Scottsdale). The students will either participate in traditional education (N=20) as is currently taking place or traditional education plus cadaver-based/simulation-based learning (N=20). Third-year medical students rotating in OB-GYN or surgery will be eligible to enroll.

Anticipated Outcomes: Knowledge-based examination results as well as performance outcomes will be improved and procedural skills and overall satisfaction will be increased.

DETAILED DESCRIPTION:
The primary goals of the final two years of medical school are to provide an experience that develops the fundamental clinical skills necessary to succeed as a resident and to offer opportunities for medical students to explore career interests. Largely unchanged for many years, the final two years of medical school include a series of required third year clerkships that include obstetrics and gynecology (OB-GYN) and general surgery. Following the completion of the third year, many students may have already decided on a specialty, and thus use the final year for electives and rotations that hone their skills and prepare them for residency. For those students planning for a procedural-based career such as OB-GYN or surgery, a considerable amount of time may be spent learning advanced surgical techniques, such as knot-tying, suturing, or other such procedures. In addition to traditional learning through didactic experiences, texts, and 'hands-on' patient interaction, some programs have developed supplemental curricula using simulators and cadaveric dissection. While studies demonstrate that these methods enhance students' readiness for procedural-based residencies, these studies have only focused on surgical residents or select fourth-year medical students who have a specific interest in surgery.

No study has focused on a comprehensive, streamlined approach using these supplemental techniques for third-year medical students. A standardized curriculum using simulation and cadaveric laboratories in the third year may provide students with the necessary skills to succeed in their required OB-GYN and surgical clerkships, while hopefully improving their examination scores and overall experience. The investigators intend to utilize a 'hands-on' series of laboratory experiences using the simulation center and cadavers to enhance the traditional learning structure. The investigators believe that a two-day course design would provide the necessary information and experience without the use of excessive resources.

Typically, work using cadavers is relegated to the study of gross human anatomy in the first year of medical school. Students experience an in-depth review of human anatomy, while learning the basic skills for dissection. After the completion of this introductory course, few medical schools routinely use cadavers or a simulation laboratory, despite the well-documented benefits for advanced learners. The usefulness of such an experience was well demonstrated in a pilot study performed by Morgan et al, which provided an intensive 78-hour (4-week) multifaceted curriculum designed for fourth year medical students prior to entering an OB-GYN residency. The course included didactic lectures, simulation training, cadaver dissection, a knot and suture experience, and surgical procedures performed on cadavers and simulation equipment. The authors concluded that despite being time-consuming and expensive, students significantly enhanced surgical skills and readiness to begin residency. Similar results have also been demonstrated in courses focused on suturing, knot-tying, and procedure-based techniques for select fourth year students entering a surgical residency program; the intent of these courses was to enhance the necessary skills to achieve appropriate required milestones. While these elective rotation pilot programs were successful in achieving their primary outcome, the drawbacks were that they were performed in fourth year students only, relegated to a select few entering surgical fields, and were costly and time-consuming.

Accordingly, the primary goal is to utilize a comprehensive, streamlined, and cost-effective approach using simulation and cadaver experiences for all eligible third-year medical students. The investigators believe that this experience will enhance scores on the Shelf and USMLE examination and improve procedural skills and overall satisfaction while remaining inexpensive and efficient. To achieve this goal, this course will be offered while students are completing their OB-GYN or general surgery rotations, both of which are heavily procedure-based and require a similar skill set. This combined effort will also allow this course to be performed six times per year instead of up to 12 times per year, which will lower costs and lessen faculty workload. If this study proves to be successful, the hope is that this curriculum could be implemented at other medical schools. The study design is also unique because the investigators will be recruiting a large student population from a national medical school instead of having students serve as their own controls in a single-center experience. The students in this study will be randomized into one of two groups: a traditional learning experience or a traditional learning experience that also includes supplemental cadaver-based and simulation-based learning.

The primary focus of this study is to determine whether the use of a comprehensive, combined, and simplified approach of using cadavers and simulation laboratories to train third-year medical students will have a beneficial effect on student performance in the OB-GYN and surgical clerkships.

Aim 1: To determine if the combined use of a 'hands-on' cadaver and simulation laboratory course will improve performance, NBME Shelf and USMLE Step 2 examination scores, and the overall experience during the third year OB-GYN and surgical clerkships.

Aim 2: To assess whether this experience can be accomplished in an efficient, cost-effective manner that would make it generalizable to other medical school curricula.

ELIGIBILITY:
Inclusion Criteria:

* All medical students in 2nd year

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Mean shelf exam scores | 1 year
  A "shelf" exam is an exam that some medical schools purchase from the NBME that test materials presented in the third-year clerkships. For this study the rotation scores examined were for obstetrics and gynecology, and surgery.

SECONDARY OUTCOMES:
Mean grade on rotation evaluation | 1 year
  The rotation evaluation is a subjective grade by the course professor.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Shapiro, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials